CLINICAL TRIAL: NCT05639426
Title: Preventing Youth Violence Through Building Equitable Communities: An Evaluation of a Systemic Intervention
Brief Title: Preventing Youth Violence Through Building Equitable Communities
Acronym: SOAR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Alabama (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Krista Mehari, Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-454; R01MD017477 (NIH)
Record Dates: First submitted 2022-11-01; First posted 2022-12-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Suicide; Violence in Adolescence
MeSH Terms: conditions — Suicide | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Strengthening Opportunities for Achievement and Resilience (Experimental): Strengthening Opportunities for Achievement and Resilience (SOAR) is an intervention condition consisting of both Culturally-Responsive Schoolwide Positive Behavior Interventions and Supports (C-SWPBS) and Culturally Responsive Practices (CRP). It is a year-long, school-level intervention.
  Interventions: Behavioral: Culturally Responsive Practices (CRP); Behavioral: Culturally-Responsive Schoolwide Positive Behavior Interventions and Supports (C-SWPBS)

INTERVENTIONS:
Behavioral: Culturally Responsive Practices (CRP) — The CRP component of the intervention targets pedagogy, curriculum, and potential teacher biases and discriminatory behavior. This component will consist of two intensive 4-hour workshops delivered by Morton and Billingsley in each school's first intervention year as well as one-hour annual boosters (Backpacks for Success and Culturally Relevant Pedagogy). All teachers and school administrators will participate in the workshops. The purpose of Backpacks for Success is to increase participants' awareness of structural racism, empathy for students, and motivation to change, while identifying equity targets and strategies to reach those targets. Culturally Relevant Pedagogy comprises classroom based strategies to promote equity, including use of culturally responsive curriculum, language, attitudes, and actions, with the goal of reducing interpersonal and cultural racism. Ongoing group coaching sessions will provide a space for peer support and learning around increasing CRP.
Behavioral: Culturally-Responsive Schoolwide Positive Behavior Interventions and Supports (C-SWPBS) — We will implement SWPBS according to the equity-focused framework established by the Center on PBIS, with an increased emphasis on community integration. SWPBS involves creating a school team of 6-10 people, including at least one administrator, teachers, and staff members. We will include at least three community stakeholders on each C-SWPBS team to integrate the culture of the community, reducing institutional and cultural racism. Community stakeholders may be parents or other invested members of the local community not employed by the school district. The school climate specialists serve on the C-SWPBS team and provide consultation for the management of violence incidents and mental health concerns.

SUMMARY:
Interpersonal or community violence is a long-standing health disparity that disproportionately affects African American youth, and suicide is disproportionately increasing among African American youth. This project evaluates the impact of a multisystemic prevention program designed to reduce health disparities in violence by promoting equity in African American youths' experiences in education systems. This intervention has the potential to reduce morbidity and mortality among African American youth, promote overall quality of life, and reduce the societal costs associated with both interpersonal violence and suicidality.

DETAILED DESCRIPTION:
Violence disproportionately affects African American youth. In addition to death and injury, violence exposure has significant psychological consequences, including traumatic stress symptoms and internalizing problems. Self-directed violence has shown startling and disproportionate growth among African American youth, with suicide rates nearly doubling from 2007 to 2018. Current prevention strategies have limited effectiveness, perhaps due to their failure to address the causal role of structural racism in violence. The primary aim of this proposed project is to examine the extent to which an intervention addressing structural racism in education reduces interpersonal violence and suicide among middle school-aged youth, with a focus on populations experiencing health disparities (African Americans; low-income communities). The proposed project will examine community-level changes using a multiple baseline experimental design that randomizes the start of the intervention in four communities, each comprising a police precinct and middle school. The intervention will consist of school-based intervention components including a culturally responsive, community-inclusive adaptation of a whole-school climate intervention (School-wide Positive Behavior Interventions and Supports) and culturally responsive practices training and coaching. Outcomes will be measured using archival data from the schools as well as survey data from youth and school personnel. Aim 1 is to evaluate the extent to which targeting structural and cultural racism reduces interpersonal violence among youth, as measured by individual-level and school-level data. Aim 2 is to evaluate the extent to which targeting structural and cultural racism reduces suicidality among youth, as measured by completed suicides and proximal precedents for suicide, including attempts and ideation. Aim 3 is to evaluate the extent to which targeting structural and cultural racism reduces both overall rates and disproportionality of school-based exclusionary discipline practices and increases culturally relevant pedagogy. Aim 4 is to evaluate specific intervention components by determining their effects on hypothesized mechanisms of change at the individual, teacher, and school levels. This intervention has the potential to reduce morbidity and mortality among African American youth, promote overall quality of life, and reduce the societal costs associated with both interpersonal violence and suicidality. Furthermore, effective strategies to address structural racism have the potential to facilitate groundbreaking public health prevention of health disparities.

ELIGIBILITY:
Inclusion Criteria:

* Youth will be eligible for the study if they attend a participating school, are capable of providing assent, and are able to understand spoken or written English.
* School personnel will be eligible if they are currently employed at a participating school.

Exclusion Criteria:

* Unable to give assent or consent.

Ages: 10 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1672 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Change in youth self-reported interpersonal violence perpetration | Trajectories of change will be assessed through data collected every three months from August to May (the school year) over the course of five years (through study completion)
  A random sample of youth will complete surveys every three months over the school year for the entire project period. To assess interpersonal violence perpetration, youth will complete the Problem Behavior Frequency Scales- Adolescent Revised, Physical Aggression subscale. Youth self-report will be aggregated to the community level to assess trajectories of community-level change over time as part of the multiple baseline design.
Change in teacher-reported youth interpersonal violence perpetration | Trajectories of change will be assessed through data collected every three months from August to May (the school year) over the course of five years (through study completion)
  Teachers will complete surveys on a random sample of youth every three months over the school year for the entire project period. To assess youth interpersonal violence perpetration, teachers will complete the Problem Behavior Frequency Scales - Teacher Report, Physical Aggression subscale. Teacher report of youth will be aggregated to the community level to assess trajectories of community-level change over time as part of the multiple baseline design.
Change in school discipline incidents for violent behavior | Trajectories of change will be assessed through data collected every three months from August to May (the school year) over the course of five years (through study completion)
  We will collect archival data from the school system by participating school and quantify the number of violence-related discipline incidents (office discipline referrals, suspensions, and expulsions) that occur every three months. Violence-related discipline incidents will be aggregated to the community level to assess trajectories in community-level change over time as part of the multiple baseline design.
Change in youth self-reported interpersonal violence victimization | Trajectories of change will be assessed through data collected every three months from August to May (the school year) over the course of five years (through study completion)
  A random sample of youth will complete surveys every three months over the school year for the entire project period. To assess interpersonal violence perpetration, youth will complete the Problem Behavior Frequency Scales- Adolescent Revised, Physical Victimization subscale. Youth self-report will be aggregated to the community level to assess trajectories of community-level change over time as part of the multiple baseline design.
Change in youth self-reported exposure to community violence | Trajectories of change will be assessed through data collected every three months from August to May (the school year) over the course of five years (through study completion)
  A random sample of youth will complete surveys every three months over the school year for the entire project period. To assess exposure to community violence, youth will complete the Survey of Children's Exposure to Violence scale. Youth self-report will be aggregated to the community level to assess trajectories of community-level change over time as part of the multiple baseline design.
Change in teacher-reported youth interpersonal violence victimization | Trajectories of change will be assessed through data collected every three months from August to May (the school year) over the course of five years (through study completion)
  Teachers will complete surveys on a random sample of youth every three months over the school year for the entire project period. To assess youth interpersonal violence perpetration, teachers will complete the Problem Behavior Frequency Scales - Teacher Report, Victimization subscale. Teacher report of youth will be aggregated to the community level to assess trajectories of community-level change over time as part of the multiple baseline design.
Change in youth self-reported suicide attempts | Trajectories of change will be assessed through data collected every three months from August to May (the school year) over the course of five years (through study completion)
  A random sample of youth will complete surveys every three months over the school year for the entire project period. To assess suicide attempts and plans, youth will complete three items from the Youth Risk Behavior Surveillance Survey, which will be summed to create a suicide attempts/plans index. Youth self-report will be aggregated to the community level to assess trajectories of community-level change over time as part of the multiple baseline design.
Change in youth self-reported suicide capacity | Trajectories of change will be assessed through data collected every three months from August to May (the school year) over the course of five years (through study completion)
  A random sample of youth will complete surveys every three months over the school year for the entire project period. To assess suicide capacity, youth will complete the Suicide Capacity Scale. Youth self-report will be aggregated to the community level to assess trajectories of community-level change over time as part of the multiple baseline design.
Change in youth self-reported suicide ideation | Trajectories of change will be assessed through data collected every three months from August to May (the school year) over the course of five years (through study completion)
  A random sample of youth will complete surveys every three months over the school year for the entire project period. To assess suicide ideation, youth will complete the suicide subscale of the Mood and Feelings Questionnaire. Youth self-report will be aggregated to the community level to assess trajectories of community-level change over time as part of the multiple baseline design.
Change in school-reported youth suicide-related incidents | Trajectories of change will be assessed through data collected every three months from August to May (the school year) over the course of five years (through study completion)
  We will collect archival data from the each participating school and quantify the number of youth suicide-related incidents based on suicide protocols administered by the school counselor every three months. Youth suicide-related incidents will be aggregated to the community level to assess trajectories in community-level change over time as part of the multiple baseline design.
Change in youth-reported race-based discrimination experiences | Trajectories of change will be assessed through data collected every three months from August to May (the school year) over the course of five years (through study completion)
  A random sample of youth will complete surveys every three months over the school year for the entire project period. To assess perceived racial discrimination, youth will complete the Adolescent Discrimination Distress Index. Youth self-report will be aggregated to the community level to assess trajectories of community-level change over time as part of the multiple baseline design.
Change in youth-reported perceptions of police | Trajectories of change will be assessed through data collected every three months from August to May (the school year) over the course of five years (through study completion)
  A random sample of youth will complete surveys every three months over the school year for the entire project period. To assess their perceptions of police legitimacy, youth will complete the Perceptions of Police scale. Youth self-report will be aggregated to the community level to assess trajectories of community-level change over time as part of the multiple baseline design.
Change in inclusive pedagogy | Trajectories of change will be assessed through data collected every three months from August to May (the school year) over the course of five years (through study completion)
  Participating teachers in each school will provide example lesson plans on every three months. These lesson plans will be coded by trained graduate students in education using the Rubric for Culturally Responsive Lessons and Assignments, which will result in an inclusive pedagogy score. These scores will be aggregated to the community level to assess trajectories in community-level change over time as part of the multiple baseline design.
Change in base rates in exclusionary discipline | Trajectories of change will be assessed through data collected every three months from August to May (the school year) over the course of five years (through study completion)
  We will collect archival data from the school system by participating school and quantify the number of exclusionary discipline incidents (a combined measure of suspensions and expulsions) that occur every three months. Exclusionary discipline incidents will be aggregated to the community level to assess trajectories in community-level change over time as part of the multiple baseline design.
Change in racial disparities in exclusionary discipline | Trajectories of change will be assessed through data collected every three months from August to May (the school year) over the course of five years (through study completion)
  We will collect archival data from the school system by participating school and quantify the number of exclusionary discipline incidents (a combined measure of suspensions and expulsions) for Black youth and White youth that occur every three months. We will use that data to create an indicator of disproportionate exclusionary discipline based on the number of exclusionary discipline events per Black youth and per White youth separately in proportion to the number of White youth and Black youth in the school. Exclusionary discipline disproportionality will be aggregated to the community level to assess trajectories in community-level change over time as part of the multiple baseline design.

SECONDARY OUTCOMES:
Change in youth self-reported traumatic stress symptoms | Trajectories of change will be assessed through data collected every three months from August to May (the school year) over the course of five years (through study completion)
  A random sample of youth will complete surveys every three months over the school year for the entire project period. To assess symptoms of posttraumatic stress disorder, youth will complete the Checklist of Children's Distress. Youth self-report will be aggregated to the community level to assess trajectories in community-level change over time as part of the multiple baseline design.
Change in youth self-reported depressive symptoms | Trajectories of change will be assessed through data collected every three months from August to May (the school year) over the course of five years (through study completion)
  A random sample of youth will complete surveys every three months over the school year for the entire project period. To assess symptoms of depression, youth will complete the Short Mood and Feelings Questionnaire. Youth self-report will be aggregated to the community level to assess trajectories of community-level change over time as part of the multiple baseline design.
Change in youth self-reported general internalizing symptoms | Trajectories of change will be assessed through data collected every three months from August to May (the school year) over the course of five years (through study completion)
  A random sample of youth will complete surveys every three months over the school year for the entire project period. To assess internalizing symptoms, youth will complete the Emotional Problems subscale of the Strengths and Difficulties Questionnaire. Youth self-report will be aggregated to the community level to assess trajectories of community-level change over time as part of the multiple baseline design.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Alabama, Mobile, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Given the sensitivity of the youth data, we do not plan to make IPD available to other researchers except under specific circumstances. We will share the data on a case-by-case basis to qualified members of the research community through a Data Use Agreement and following documentation that they have obtained the approval of an institutional review board. We will ensure that all released data have appropriate documentation that describes the method of collection, what the data represent, and potential limitations for use by creating a Data Codebook. This report will include (1) documentation of the measures and evidence of internal validity; and (2) participant recruitment, recruitment rates, and information about the survey administration process. Data will be self-archived on a secure university network drive through the university's library system. Vanderbilt University will be responsible for long-term preservation of the data.